CLINICAL TRIAL: NCT03482401
Title: Metabolic Profiling of Dietary Polyphenols and Methylxanthines in Normal and Malignant Mammary Tissues From Breast Cancer Patients
Brief Title: Disposition of Dietary Polyphenols and Methylxanthines in Mammary Tissues From Breast Cancer Patients
Acronym: POLYSEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Council, Spain (Other Government)
Collaborators: Hospital General Universitario Reina Sofía de Murcia (Other)
Responsible Party: Principal Investigator, Juan Carlos Espín de Gea, Research Professor, National Research Council, Spain
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 201770E081
Record Dates: First submitted 2018-03-15; First posted 2018-03-29 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer
Keywords: Polyphenol; Methylxanthine; Metabolism; Breast tissue; Disposition; UPLC-QTOF
MeSH Terms: conditions — Breast Neoplasms | interventions — Polyphenols

STUDY DESIGN:
Intervention Model Description: Randomised, parallel-controlled dietary intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polyphenol group (Experimental): Patients consumed a polyphenol-rich dietary supplement (commercial lemon, orange, pomegranate, olive, grape, cocoa, curcuma and broccoli extracts), mainly rich in simple phenolics such as hydroxytyrosol and the polyphenols procyanidins, hesperidin, eriocitrin, curcumin, resveratrol, punicalagin and ellagic acid. Cocoa extract also contains the methylxanthines theobromine and caffeine.
  Interventions: Dietary Supplement: Polyphenol
- Control group (No Intervention): Participating patients did not consume the supplement but provided biological samples to the trial

INTERVENTIONS:
Dietary Supplement: Polyphenol — Patients consume 3 capsules/day (474 mg phenolics/day) from the biopsy-confirmed breast cancer diagnosis to the surgery
  Arms: Polyphenol group

SUMMARY:
The aim is to characterise the metabolic profiling of dietary polyphenols in normal and malignant breast tissues from breast cancer patients.

DETAILED DESCRIPTION:
The objective of this exploratory trial is to determine the disposition and characterise the metabolic profiling of dietary polyphenols in normal and malignant glandular breast tissues from newly diagnosed breast cancer patients.

The patients consumed a polyphenol-rich dietary supplement containing 37 different phenolics and 2 methylxanthines (theobromine and caffeine) from the diagnosis to the surgery. The metabolic profiling was characterized in normal and malignant breast tissues as well as plasma and urine using UPLC-ESI-QTOF-MS/MS.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients are those over 18 years with a newly biopsy-confirmed breast cancer, programmed surgery at least 3 days after the recruitment and no neoadjuvant treatment.

Exclusion Criteria:

* Suspected intolerance to any component of fruits or vegetables.
* Neoadjuvant chemo- or radiotherapy.
* Urgent surgery (less than 3 days after the recruitment).
* Patient under 18 years.
* Patient with breast adenoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Quantification of dietary polyphenols and methylxanthines in breast tissues | 1-24 months
  Quantification of dietary polyphenols and methylxanthines in normal and malignant mammary tissues from breast cancer patients using ultra-high resolution liquid chromatography coupled to quadrupole-time-of-flight mass spectrometry (UPLC-ESI-QTOF-MS/MS).
  * Quantification (pmol/g) of each phenolic-derived metabolite in breast tissues.
  * Quantification (pmol/g) of each methylxanthine-derived metabolite in breast tissues.

SECONDARY OUTCOMES:
Quantification of dietary polyphenols and methylxanthines in plasma and urine | 8-24 months
  Quantification of dietary polyphenols and methylxanthines in urine and plasma from breast cancer patients using ultra-high resolution liquid chromatography coupled to quadrupole-time-of-flight mass spectrometry (UPLC-ESI-QTOF-MS/MS).
  * Quantification of each phenolic-derived metabolite in urine and plasma (nmol/L).
  * Quantification of each methylxanthine-derived metabolite in urine and plasma (nmol/L).

CONTACTS AND LOCATIONS:
Overall Officials: Juan C. Espín, PhD, Principal Investigator — National Research Council, Spain
Locations (1):
- Hospital General Universitario Reina Sofía, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No